CLINICAL TRIAL: NCT01463176
Title: Music Therapy as Procedural Support for Young Children Undergoing Immunizations: A Randomized Controlled Study
Brief Title: Music Therapy as Procedural Support for Young Children Undergoing Immunizations
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Florida State University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 2011.6797
Record Dates: First submitted 2011-10-20; First posted 2011-11-01 (Estimated); Last update posted 2015-08-11 (Estimated); Status verified 2015-08

CONDITIONS: Immunization
Keywords: Music Therapy; Child Psychology; Vaccination
MeSH Terms: interventions — Music Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Standard Care (No Intervention): Children in the Standard Care Control group will receive standard care and will be videotaped by the music therapist but will not receive music therapy during their immunization
- Music Therapy (Experimental): Children in this group will receive live music therapy during their immunization.
  Interventions: Behavioral: Music Therapy

INTERVENTIONS:
Behavioral: Music Therapy — Live music therapy is interactive and incorporates behavioral cues for coping techniques during the procedure, using patient-preferred music.
  Arms: Music Therapy

SUMMARY:
Many young children undergo medical procedures that are painful and distressing. Negative experiences during medical procedures can have serious long-term effects, including fear and avoidance of medical procedures during adulthood. Distraction interventions can help prevent children from forming negative memories of medical procedures. Live music therapy has been shown to alleviate pediatric distress during both invasive and non-invasive procedures. The objective of this study is to examine the effects of music therapy on the child's distress behaviors and time to calm, as well as the length of the procedure and use of restraint, and parents' and healthcare staffs' behaviors during the procedure, for young children undergoing immunizations and influenza vaccinations. It is hypothesized that children receiving music therapy will show fewer distress behaviors, calm more quickly, and have shorter procedures with fewer instances of restraint compared to children who receive standard care. In addition, it is predicted that adults (parents and staff) will show fewer distress-promoting behaviors during, before, and after the procedures.

ELIGIBILITY:
Inclusion Criteria:

* Participants will be pediatric patients (N = 60) from 48 to 72 months of age who are undergoing immunizations, as well as their parents/legal guardians (N = 60) and the healthcare staff who are conducting/assisting with their procedure (N = 60).

Exclusion Criteria:

* Any children whose parents are non-English speakers or staff who are non-English speakers will be excluded.

Ages: 48 Months to 72 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 150 (Actual)
Dates: Start 2011-10; Primary Completion 2012-08 (Actual); Study Completion 2012-08 (Actual)

PRIMARY OUTCOMES:
Child's behavioral distress, as measured by the Children's Hospital of Eastern Ontario Pain Scale (CHEOPS) | From the time the nurse enters the treatment room until the child leaves the treatment room after the procedure (approximately 5-10 minutes)
  Distress will be assessed at fifteen second intervals throughout the procedure by trained observers upon review of videos of procedures (within approximately one month of procedure)

SECONDARY OUTCOMES:
Child and adult behaviors, as measured by the Child-Adult Medical Procedure Interaction Scale- Short Form (CAMPIS-SF) | From the time the nurse enters the treatment room until the child leaves the treatment room after the procedure (approximately 5-10 minutes)
  Child and adult behaviors will be assessed at fifteen second intervals throughout the procedure by trained observers upon review of videos of procedures (within approximately one month of procedure).
Child's pain and distress, reported by the child's parent using the Universal Pain Assessment Tool | After the procedure, when the child and parent have left the treatment room (within approximately 5 minutes of the procedure).
Parent perceptions of and satisfaction with the procedure, measured using a researcher-designed satisfaction survey | After the procedure, when the child and parent have left the treatment room (within approximately 5 minutes of the procedure).
Length of time it takes the child to calm after the procedure, in minutes and seconds | Observers will begin recording the length of time to calm starting with the needle insertion and ending when the child receives a CHEOPS score of 6 or less (within approximately 5 minutes after needle insertion).
  Assessed by trained observers upon review of a video tape of the procedure (within approximately a month of the procedure)

CONTACTS AND LOCATIONS:
Overall Officials: Olivia S Yinger, MME, Principal Investigator — Florida State University
Locations (3):
- United States (3):
  - Tallahassee Primary Care Associates, Tallahassee, Florida
  - Tallahassee Memorial HealthCare Family Medicine Clinic, Tallahassee, Florida
  - Memorial Pediatrics, Bainbridge, Georgia